CLINICAL TRIAL: NCT03727737
Title: Efficacy of Repetitive Transcranial Magnetic Stimulation for Improvement of Memory in Older Adults With TBI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: Stanford University (Other); The Defense and Veterans Brain Injury Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Maheen M Adamson, Senior Scientific Research Director, Defense and Veterans Brain Injury Center (DVBIC), Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ADA0007AGG
Record Dates: First submitted 2018-10-23; First posted 2018-11-01 (Actual); Last update posted 2023-04-11 (Actual); Status verified 2023-04

CONDITIONS: Brain Injuries, Traumatic; Repetitive Transcranial Magnetic Stimulation; Memory Deficits; Aging
Keywords: repetitive Transcranial Magnetic Stimulation; Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic; Memory Disorders | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The proposed study will evaluate the safety, durability and efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) as a promising non-invasive therapeutic treatment for improving memory in older adults with mild or moderate Traumatic Brain Injury (TBI) who have been experiencing residual memory or cognitive problems that affect daily functioning.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind study until trial is complete
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham (No Intervention): Patients with mild and moderate TBI will be assigned randomly to this arm and will not receive treatment
- ACTIVE (Active Comparator): Patients with mild and moderate TBI will be assigned randomly to this arm and will receive treatment
  Interventions: Device: Repetitive Transcranial magnetic Stimulation

INTERVENTIONS:
Device: Repetitive Transcranial magnetic Stimulation — RTMS will be delivered via magventure machine, on an approved FDA IDE protocol to DLPFC region to improve memory in older adults (veterans and non-veterans) with mild and moderate TBI.
  Other Names: rTMS
  Arms: ACTIVE

SUMMARY:
The proposed study will evaluate the safety, durability and efficacy of repetitive Transcranial Magnetic Stimulation (rTMS) as a promising non-invasive therapeutic treatment for improving memory in older adults with mild or moderate Traumatic Brain Injury (TBI) who have been experiencing residual memory or cognitive problems that affect daily functioning.

DETAILED DESCRIPTION:
Recent advances in both AD and TBI test non-pharmaceutical interventions that target chronic symptom improvement (e.g., non- invasive brain stimulation, exercise and cognitive training). In order to provide targeted therapies to patients who suffer from chronic sequela of TBI it is necessary to understand mechanisms of repair within the context of an aging brain. Repetitive TMS (rTMS) delivers therapeutic, noninvasive brain stimulation, is FDA-approved for treatment for major depression and currently used for treatment of pain, PTSD, anxiety, improvement of executive function in mild and moderate TBI, severe TBI, memory enhancement and dementia.

This treatment can induce neuronal long-term potentiation resulting in synaptic repair leading to improvements in memory function through hippocampal- cortical circuits and brain connectivity measured by resting state-fMRI (rs fMRI) particularly in default mode and central executive network (DMN & CEN). The study primarily proposes to assess the efficacy of rTMS to improve memory performance and to test rs-fMRI (i.e. DMN) as a potential biomarker to capture response to treatment in older patients suffering with chronic symptoms related to previous brain injuries (depression, PTSD etc). In addition, the study will assess other established biomarkers longitudinally (e.g.,hypometabolism via PET FDG, cortical oscillation via electroencephalography (EEG), Brain Derived Nerve Growth Factor (BDNF)and hippocampal volume from structural MRI) to capture patient response to treatment that may signal early dementia.

HYPOTHESES:

Primary:

Subjects with TBI who receive active rTMS treatment (rTMS_A) will: a) show significantly greater improvement from baseline in memory performance post rTMS intervention compared to subjects who received sham rTMS treatment (rTMS_S), and b) show stronger functional connectivity within and between DMN and CEN post rTMS intervention compared to patients who received sham (rTMS_S).

Secondary:

1. Quality of Life (QOL): scores on QOL scale will improve with rTMS treatment in patients who receive rTMS treatment.
2. Sustained Improvement: At 6-month follow-up, patients with TBI in rTMS_A group would be more likely to have sustained greater brain connectivity compared to patients in the rTMS_S group predicting better memory performance.
3. Moderators of Response: The following variables may moderate memory function improvement in patients with TBI post intervention and at 6-month follow-up: Age, health condition variables (severity of symptoms at baseline, time to injury, baseline cognitive performance, TBI type,comorbidities (PTSD, sleep, depression), substance abuse, medication use, fatigue); physiological and biological variables (baseline hippocampal volume and/or microstructure, baseline connectivity in DMN & CEN, EEG resting and task-related cortical oscillations, and Brain Derived Neurotrophic Factor (BDNF) genotype.
4. Mediators of Response: To assess the mechanism of rTMS in synaptic repair/regeneration, pre and post changes will be assessed in depression and PTSD measures, Plasma BDNF, FDG PET hypometabolism in precuneus/posterior cingulate area, EEG resting and task-related cortical oscillations, and connectivity of DLPFC (stimulation site & part of CEN) with other DMN.

SPECIFIC OBJECTIVES:

Primary Objective: a) To assess the efficacy of rTMS to predict improvement in memory performance pre and post rTMS intervention in older patients with TBI, and b) To assess rs-fMRI as a biomarker to detect these changes in memory performance.

Secondary Objective: To assess the mechanism of rTMS in synaptic repair/regeneration by assessment of structure & functional brain activity (PET/MRI, fMRI, & EEG), genetic, cognitive and behavioral function factors (including QOL, depression and PTSD).

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years, with a high school education
* History of mild or moderate TBI as defined by the DoD/VA Clinical Practice Guidelines for Definition of TBI
* Ability to obtain a Motor Threshold (MT) will be determined during the screening process
* Must be in the chronic stable phase of recovery (>6 months post injury) with residual cognitive difficulties that are affecting daily functioning (including self-reported memory or cognition problems)
* If on a psychotropic medication regimen, that regimen will be stable for at least 4 weeks prior to entry to the study and patient will be willing to remain on a stable regimen during the acute treatment phase
* Has an adequately stable condition and environment to enable attendance at scheduled clinic visits
* For female participants of child bearing potential, agrees to use one of the following acceptable methods of birth control: abstinence, oral contraceptive, Norplant, Depo-Provera, a condom with spermicide, a cervical cap with spermicide, a diaphragm with spermicide, an intrauterine device, surgical sterilization (having your tubes tied)
* Able to read, verbalize understanding, and voluntarily sign the Informed Consent Form prior to participating in any study-specific procedures or assessments
* Individuals who meet the study criteria but have impaired decision making capacity may participate provided they are able to voluntarily sign an Assent Form and have an LAR who can sign a Consent Form and accompany the participant to all study visits

Exclusion Criteria:

* Diagnosed with Dementia
* Pregnant or lactating female.
* Unable to be safely withdrawn, at least two-weeks prior to beginning treatment, from medications that substantially increase the risk of seizures
* Have a cardiac pacemaker or a cochlear implant
* Have an implanted device (deep brain stimulation) or metal in the brain (see standard MRI exclusion criteria including metal screening section in telephone screen, Appendix A)
* Have a mass lesion, cerebral infarct or other active CNS disease, including a seizure disorder
* Known current psychosis as determined by DSM-IV coding in chart (Axis I, psychotic disorder, schizophrenia) or a history of a non-mood psychotic disorder
* Diagnosis of Bipolar Affective Disorder I (as determined by chart review and intake interview), since this in conjunction with TBI increases seizure risk
* Current amnesic disorders, dementia, MOCA ≤ 16, or delirium.
* Current substance abuse (not including caffeine or nicotine) as determined by positive toxicology screen, or by history via AUDIT, within 3 months prior to screening
* Prior history of seizures
* Severe TBI or open head injury
* TBI within last 6 months
* Participation in another concurrent clinical trial
* Patients with prior exposure to rTMS (NOTE: TMS is allowed) or ECT
* Active current suicidal intent or plan. Patients at risk for suicide will be required to establish a written safety plan involving their primary psychiatrist. All patients at risk for suicide will be excluded from the study (as per FDA recommendation).

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-23 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2022-09-14 (Actual)

PRIMARY OUTCOMES:
CANTAB Paired Associates Learning (PAL) | 2-4 weeks
  Test for visual memory and new learning: it is a hippocampal-mediated paired associates learning task. This test has twenty-one outcome measures, covering the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed (Administration time 10 minutes). The main score provided is the sum of pairs reproduced over three trials (range: 0-30). We will use the average number of trials needed to succeed on PAL task as the main outcome measure.

SECONDARY OUTCOMES:
Functional Connectivity Changes in the Brain | 2-4 weeks
  Neuroimaging using PET/MRI to determine Functional Connectivity in Default Mode Network (DMN) and Central Executive Network (CEN) systems in the brain following rTMS treatment. we will do this by doing ICA analysis for each network focused from the stimulation site.

OTHER OUTCOMES:
Quality of Life measure: Short Form of Veterans Rand 36 Item Health Survey (SF/VR-36) | 2-4 weeks
  Measure of Quality of Life change following rTMS treatment. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability. We will look at these standardized eight scores as outcomes measures as well as a total composite score as an outcome measure.
Sustained Improvement in primary Outcome Measure (CANTAB Paired Associates Learning (PAL)) at 6 months post-treatment | 6 months
  At 6-month follow-up, the study primary outcome, CANTAB Paired Associate Learning task will be assessed again to identify changes that are sustained due to treatment at six-months. This test has twenty-one outcome measures, covering the errors made by the participant, the number of trials required to locate the pattern(s) correctly, memory scores and stages completed (Administration time 10 minutes). The main score provided is the sum of pairs reproduced over three trials (range: 0-30). We will use the average number of trials needed to succeed on PAL task as the main outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States